CLINICAL TRIAL: NCT03445676
Title: Multi-center, Randomized Non-inferiority Trial to Determine if Using Alcohol-based Hand Rub to Clean Gloved Hands When an Indication for HH Arises During a Single Patient Encounter is as Effective as Current Recommendation and Standard Care
Brief Title: Effectiveness of an Alcohol-based Hand Rub to "Clean" Gloved Hands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kerri A Thom, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00065976/69543
Record Dates: First submitted 2018-02-06; First posted 2018-02-26 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Hand Hygiene
Keywords: Hand Hygiene; WHO 5-moments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Study personnel silently observe and record what the healthcare worker does at each hand hygiene opportunity without direction to the healthcare worker
- ABHR directly on gloves (Experimental): Healthcare worker will be directed by study personnel to use alcohol-based hand rub (ABHR) to cleanse gloves at each hand hygiene opportunity
  Interventions: Behavioral: ABHR directly on gloves
- Ideal Standard (Placebo Comparator): Healthcare worker will be directed by study personnel to remove gloves, perform hand hygiene and replace gloves at each hand hygiene opportunity
  Interventions: Behavioral: ABHR directly on gloves

INTERVENTIONS:
Behavioral: ABHR directly on gloves — HCW will be directed by study personnel to use alcohol-based hand rub (ABHR) to cleanse gloves at each hand hygiene opportunity
  Arms: ABHR directly on gloves; Ideal Standard

SUMMARY:
Although little is known about compliance with the World Health Organization (WHO) 5 Moments of hand hygiene, the few existing studies report a high number of opportunities and compliance ranging from just 22 to 60%. Previous studies have reported an increased density of opportunities, perceived insufficient time and glove use as factors associated with non-compliance. A healthcare worker performing multiple tasks in one encounter may spend up to half the time in the room doing hand hygiene. Strategies to reduce the time required for hand hygiene may in turn promote increased compliance and may ultimately be most effective in limiting microbial transmission. In this study, the investigators examine whether cleansing gloves at each hand hygiene opportunity at the point of care and reusing the same gloves is as effective as standard practice and the current recommendation (remove gloves, perform hand hygiene, and don new gloves).

DETAILED DESCRIPTION:
During this multi-center, randomized non-inferiority trial, eligible healthcare personnel entering rooms of patients on Contact Precautions (or other rooms in which hand hygiene (HH) is an expectation) and who agree to study participation will be randomized to either ideal standard (healthcare worker (HCW) will be directed by study personnel to remove gloves, perform hand hygiene and replace gloves at each HH opportunity), experimental glove-reuse (HCW will be directed by study personnel to use alcohol-based hand rub (ABHR) to cleanse gloves at each HH opportunity) or usual care (study personnel silently observe and record what the HCW does at each HH opportunity without direction to the HCW).Care for patients with C. difficile will be excluded as ABHR is not recommended.

This study will be performed at the University of Maryland Medical Center, The R.Adams Cowley Shock Trauma Hospital, University of Iowa Hospitals and The Johns Hopkins Hospital. Healthcare workers on any patient units will be potentially eligible, but the investigators will strive for diversity across unit types (e.g. adult med-surg, general pediatrics, adult ICUs, emergency care areas and inpatient hemodialysis units). The investigators will use a stratified, block randomization scheme to ensure an equal number of participants from each participating unit and facility. The HCW, regardless of random assignment, may choose to remove gloves at any point (e.g. if gloves are heavily soiled or are compromised).

All participants will be instructed on how to perform HH using the standardized WHO methodology and will also receive brief instruction regarding HH opportunities at the point of care using a WHO 5 Moments pamphlet. Participants will don gloves and enter the room to perform patient care activities as planned. Research staff will be in the room to monitor the HCW activity. Research staff trained using the WHO Hand Hygiene Monitoring Method will identify HH opportunities. At each opportunity, the participant will be instructed to stop current activity in the intervention and ideal standard group. Participants in the intervention group will be instructed to cleanse gloves using an ABHR in a standardized way and in a similar fashion to the WHO recommendations for HH. Participants in the ideal standard group will be instructed to remove gloves, perform HH using an ABHR, and don new gloves. The HCW will continue with planned activities and continue to cleanse gloves or perform HH according to study assignment for each opportunity until either the HCW has completed patient care or five HH events have occurred. Study staff will record what the HCW randomized into the usual care arm does at each HH moment. The investigators chose a maximum of five HH events because since most encounters will have five or fewer HH opportunities.

After the final opportunity and after cleansing gloves and allowing them to dry (Intervention Group, glove reuse) after donning new gloves (Ideal Standard) or at moment 5 or before room exit which ever comes first (Usual Care Group) the non-dominant gloved hand will be sampled by directly imprinting the non-dominant gloved hand onto an agar plate. HCWs who have no HH opportunities while at the point of care (e.g. a nurse who enters to the room and interacts only with the intravenous pump and performs HH at exit) will be withdrawn from the study

ELIGIBILITY:
Inclusion Criteria:

* Healthcare worker who directly interacts with patients on Contact Precautions

Exclusion Criteria:

* Adults <18 years of age
* Care for patients with known C. difficile infection
* No hand hygiene opportunities while at the point of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1450 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Total bacteria colony forming units | Through study completion,about 1 year
  Total bacterial colony forming units cultured from gloved hands will be compared between the intervention and usual care group and between the intervention and ideal standard using a comparison of proportions.

SECONDARY OUTCOMES:
Presence of pathogenic organisms | Through study completion,about 1 year
  The presence of pathogenic bacteria on gloved hands in each arm during a single patient encounter

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Thom, MD, Principal Investigator — University of Maryland, College Park
Locations (3):
- United States (3):
  - University of Iowa Hospitals, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thom KA, Rock C, Robinson GL, Reisinger HRS, Baloh J, Chasco E, Liang Y, Li S, Diekema DJ, Herwaldt LA, Johnson JK, Harris AD, Perencevich EN. Alcohol-based decontamination of gloved hands: A randomized controlled trial. Infect Control Hosp Epidemiol. 2024 Apr;45(4):467-473. doi: 10.1017/ice.2023.243. Epub 2023 Nov 23. PMID 37994538